CLINICAL TRIAL: NCT05465291
Title: Effect of Neuromuscular Electrical Stimulation and Early Physical Activity on ICU Acquired Muscle Weakness in Mechanically Ventilated Patient: A Randomized Controlled Trial
Brief Title: Neuromuscular Electrical Stimulation in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sahar Younes, Assistant professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Neuromuscular stimulation
Record Dates: First submitted 2022-07-06; First posted 2022-07-19 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Neuromuscular Electrical Stimulation; ICU Acquired Muscle Weakness
Keywords: Mechanical ventilation; Rehabilitation; Critical care; Physiotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional care (No Intervention): Control Group
- Exercise Group (Experimental): Passive/active range of motion exercises group
  Interventions: Procedure: Exercise group
- Neuromuscular Electrical Muscle Stimulation group (Experimental): Neuromuscular Electrical Muscle Stimulation group
  Interventions: Procedure: Neuromuscular Electrical Muscle Stimulation group
- Combined therapy (Neuromuscular Electrical Muscle Stimulation pulse limb exercise) (Experimental): Combined therapy (Neuromuscular Electrical Muscle Stimulation pulse limb exercise).
  Interventions: Procedure: Neuromuscular Electrical Muscle Stimulation and Exercise group

INTERVENTIONS:
Procedure: Exercise group — This group will receive passive/active range of motion (ROM) exercises. ROM exercises will include major muscle groups (i.e. biceps, triceps, and lower limbs) and will be applied from second day till seventh day of admission .
  Other Names: EX Group
  Arms: Exercise Group
Procedure: Neuromuscular Electrical Muscle Stimulation group — * Patients in NEMS group will receive neuromuscular electrical stimulation from second day till seventh day of admission.
  * Neuromuscular electrical stimulation will be implemented simultaneously on the rectus femoris, vastus lateralis, and vastus medialis muscles of both lower limbs, with two stimulators, in two 30-min sessions per day starting from the second day till seventh day of admission .
  Other Names: NEMS group
  Arms: Neuromuscular Electrical Muscle Stimulation group
Procedure: Neuromuscular Electrical Muscle Stimulation and Exercise group — Patients in this group will be subjected to Neuromuscular Electrical Muscle Stimulation and Exercise.
  Other Names: NMES + EX group
  Arms: Combined therapy (Neuromuscular Electrical Muscle Stimulation pulse limb exercise)

SUMMARY:
Intensive care unit-acquired muscle weakness (ICUAMW) is a common problem following an ICU admission and is associated with prolonged hospitalization, delayed weaning and increased mortality. Up to 25% of patients requiring mechanical ventilation (MV) for greater than 7 days develop ICUAW, and this figure may rise to 50-100% in the septic population. Long-term follow-up studies of survivors of critical illness have demonstrated significantly impaired health-related quality of life and physical functioning up to 5 years after ICU discharge, with weakness being the most commonly reported physical limitation. Early rehabilitation has been shown to be safe and feasible; however, commencement is often delayed due to a patient's inability to cooperate. An intervention that begins early in ICU admission without the need for patient volition may be beneficial in attenuating muscle wasting. Therefore, this study aims to evaluate the effect of neuromuscular electrical stimulation and early physical activity on ICU acquired muscle weakness in mechanically ventilated patient

DETAILED DESCRIPTION:
A randomized controlled study will be carried out to achieve the aim of the current study. For three months, from July 15, 2022 to September 15, 2022, newly admitted patients will be screened. Patients in this trial will be recruited prospectively within 24 hours of admission to the general ICU. Computer-generated randomization will be used to assign patients to one of four groups: neuromuscular electrical stimulation (NMES), exercise (EX); combined therapy (NMES + EX); or conventional care (control group). A minimum total sample size of 120 samples will be included. According to sample size calculations treatment groups (NMES, EX, NMES + EX or conventional care) would be represented by a minimum of 30 patients. A total sample size a 120 will be selected for the study. All patients in the four groups will receive ICU standard care which includes sedation and weaning protocols.

Conventional care (Control Group):

Patients in this group will receive usual physiotherapy consisting of in-bed EXs and ICU standard care.

Exercise group (EX Group):

This group will receive passive/active exercise range of motion (ROM) exercises . ROM exercises will include major muscle groups (i.e. biceps, triceps, and lower limbs) and will be applied the second day of 1CU admission for seven days.

Neuromuscular Electrical Muscle Stimulation (NEMS Group):

Patients in NEMS group will receive neuromuscular electrical stimulation from the second day of ICU admission for seven days.

Neuromuscular electrical stimulation will be implemented simultaneously on the rectus femoris, vastus lateralis, and vastus medialis muscles of both lower limbs, with two stimulators, in two 30-min sessions per day starting from the second day after admission for seven days.

Combined therapy (NMES + EX):

Patients in this group will be subjected to NMES pulse EX. The application of NMES occurring simultaneously to the upper and lower limbs exercises.

The ICU acquired muscle weakness assessment tool will be developed by the researchers to assess and record occurrence of ICUAMW.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years,
* mechanically ventilated for ≥48 h
* remain in the intensive care ≥4 days.

Exclusion Criteria:

* Pre-existing neuromuscular disease
* brain death
* peripheral vascular diseases (arterial lower limb disease and deep venous thrombosis)
* hemiplegia/quadriplegia
* lower limb amputation
* spinal injuries
* receiving muscle relaxant; cognitive impairment; body mass index (BMI) > 35 kg/m2; bone fractures
* skin lesions
* presence of cardiac pacemaker
* end-stage cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
Assessing a change in limb muscle strength | on day 2 of ICU admission, on day 3, and on day 5.
  Limb muscle strength using Medical Research Council score (MRCS). Three muscle groups in all four limbs will be assessed with the MRC scale with values ranging from 0 (quadriplegia….severe muscle weakness) to 60 (normal muscle strength).

SECONDARY OUTCOMES:
Time to weaning off the ventilator | After day 2 of ICU admission and on day 5.
  Time to weaning off the ventilator
Duration of MV | After day 2 of ICU admission and on day 5.
  Duration of mechanical ventilation
ICU length of stay | After day 2 of ICU admission and on day 5.
  ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Y Othman, Assit. Prof., Principal Investigator — Faculty of Nursing, Damanhour University
Locations (1):
- Faculty of nursing, Damanhūr, Behira, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cusack R, Bates A, Mitchell K, van Willigen Z, Denehy L, Hart N, Dushianthan A, Reading I, Chorozoglou M, Sturmey G, Davey I, Grocott M. Improving physical function of patients following intensive care unit admission (EMPRESS): protocol of a randomised controlled feasibility trial. BMJ Open. 2022 Apr 15;12(4):e055285. doi: 10.1136/bmjopen-2021-055285. PMID 35428629
- [Background] McWilliams D, Weblin J, Atkins G, Bion J, Williams J, Elliott C, Whitehouse T, Snelson C. Enhancing rehabilitation of mechanically ventilated patients in the intensive care unit: a quality improvement project. J Crit Care. 2015 Feb;30(1):13-8. doi: 10.1016/j.jcrc.2014.09.018. Epub 2014 Oct 2. PMID 25316527
- [Background] Cerqueira TCF, de Cerqueira Neto ML, Cacau LAP, de Araujo Filho AA, Oliveira GU, da Silva Junior WM, Carvalho VO, de Mendonca JT, de Santana Filho VJ. Effect of neuromuscular electrical stimulation on functional exercise capacity in patients undergoing cardiac surgery: A randomized clinical trial. Clin Rehabil. 2022 Jun;36(6):789-800. doi: 10.1177/02692155211070945. Epub 2021 Dec 31. PMID 34971331
- [Background] Gomes Neto M, Oliveira FA, Reis HF, de Sousa Rodrigues- E Jr, Bittencourt HS, Oliveira Carvalho V. Effects of Neuromuscular Electrical Stimulation on Physiologic and Functional Measurements in Patients With Heart Failure: A SYSTEMATIC REVIEW WITH META-ANALYSIS. J Cardiopulm Rehabil Prev. 2016 May-Jun;36(3):157-66. doi: 10.1097/HCR.0000000000000151. PMID 26784735
- [Background] Sumin AN, Oleinik PA, Bezdenezhnykh AV, Ivanova AV. Neuromuscular electrical stimulation in early rehabilitation of patients with postoperative complications after cardiovascular surgery: A randomized controlled trial. Medicine (Baltimore). 2020 Oct 16;99(42):e22769. doi: 10.1097/MD.0000000000022769. PMID 33080746
- [Result] Burgess LC, Venugopalan L, Badger J, Street T, Alon G, Jarvis JC, Wainwright TW, Everington T, Taylor P, Swain ID. Effect of neuromuscular electrical stimulation on the recovery of people with COVID-19 admitted to the intensive care unit: A narrative review. J Rehabil Med. 2021 Mar 18;53(3):jrm00164. doi: 10.2340/16501977-2805. PMID 33634830